CLINICAL TRIAL: NCT02441647
Title: Clinical Study to Prove Safety in Use (Irritability and Sensitization in Genital Mucosa) of an Intimate Lubricating Gel
Acronym: CL STD SAF USE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kley Hertz S/A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: KLEY HERTZ-003
Record Dates: First submitted 2015-04-15; First posted 2015-05-12 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Female Dry Genital Mucosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Device: KL029 Intimate Lubricant Gel

INTERVENTIONS:
Device: KL029 Intimate Lubricant Gel

SUMMARY:
The purpose of this study is to check the safety under normal conditions of use through the emergence of signs of irritability and sensitization of the genital mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 25 to 55 years old
* Regular Menstrual Cycle
* Intact skin in product analysis área
* No prior reactions to topical products
* Being a user of products from the same category
* Reading, understanding, agreement and signature of the informed consent form

Exclusion Criteria:

* Pregnancy or risk of pregnancy
* Lactation
* Use of anti-inflammatory and immunosuppressive from 30 days up to three months prior to selection;
* Diseases that cause imune suppression;
* Endocrine disorders such as thyroid, ovarian or adrenal gland disorders;
* Any infection in the region where the product will be analyzed diagnosed at enrollment;
* Other conditions considered by the investigator physician as reasonable for the disqualification of the individual's participation in the study.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Emergence of signs of irritability and sensitization in the genital mucosa through Wilcoxon test | 40 days
  For the safety assessment, the variables will be evaluated for each experimental period using one-tailed Wilcoxon test to investigate the following hypotheses:
  H0: The median of the results of the variable under study is zero (no irritation) H1: The median of the results of the variable under study is greater than zero (no irritation) The Wilcoxon test is used because it is the ideal to compare variables collected with ordinal scale with a reference value. In this study, the reference value is zero (no irritation).
  The expectation is the absence of positive safety, ie higher scores than zero. If there are positive evidence of (mild, moderate or severe) for parameters erythema, peeling,blistering and swelling, the results are statistically evaluated.